CLINICAL TRIAL: NCT04054934
Title: Influence of Circadian Clock on Diurnal Dietary Intake, Glucose Variability, Time Spent in Range, and Neuro-cognitive Achievements Among Adolescents With and Without Type 1 Diabetes
Brief Title: Influence of Circadian Clock on Hormonal, Metabolic, Neurocognitive Markers in Adolescents With and Without Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Western University, Canada (Other); Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Head of Pediatric Endocrinology Unit, Assaf-Harofeh Medical Center
Other Study IDs: 0291-18
Record Dates: First submitted 2019-05-26; First posted 2019-08-13 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: T1DM; Sleep Disorders, Circadian Rhythm; ADHD; Memory Impairment
Keywords: T1DM; Hypothalamus; CORTICAL BRAIN; Glucose variability; Biological clock; Pediatrics
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Attention Deficit Disorder with Hyperactivity; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Circardian rhythm: Regular night sleep, with at least 7 hours length of sleep.
  Interventions: Behavioral: Normal Circadian Rhythm
- Reversed circadian rhythm: Night/day circadian clock is opposite, with at least 7 hours length of sleep
  Interventions: Behavioral: Reversed Circadian Rhythm

INTERVENTIONS:
Behavioral: Reversed Circadian Rhythm — Revered day/ night sleep cycle
  Groups: Reversed circadian rhythm
Behavioral: Normal Circadian Rhythm — Normal day/ night sleep cycle
  Groups: Normal Circardian rhythm

SUMMARY:
Type 1 diabetes mellitus (T1DM), makes its appearance during childhood and youth, but management implications last till late adulthood. Its treatment includes the combination of multiple daily glucose measurements, insulin administration and balanced nutrition. The goals of therapy are to achieve glycemic control (HbA1c < 7.5%), and minimal glycemic excursions. Furthermore, recent studies imply that keeping HbA1c within target range is not sufficient to prevent complications, attributed mainly to blood glucose level fluctuating from high to low, associated with food intake and adolescents behavior. The current implication of glycemic control on the central nervous system (CNS) includes abnormal electrical brain activity, structural changes in brain's white and grey matter, and cognitive impairment. Still, little is known on the effect of sleep pattern, including circadian rhythm reversal ("biological clock) on asymptomatic glycemic excursions, and on CNS functions. There is no data regarding the association of the biologic clock on CNS functionality among adolescents, nonetheless among T1DM adolescents, for whom behavior and circadian rhythm alterations may have harmful effect. The investigators propose a cross-over designed study by examining adolescents with and without T1DM during 2 weeks of regular sleeping pattern (night sleep), and during 2 weeks of sleeping during the day as happens during summer vacation. The main objective of the proposed study is to offer proof of the clinical and metabolic relevance and cognitive effects of the reversal of the circadian clock in adolescents with and T1DM during summer vacations and weekends. Study is designed to demonstrate a difference among healthy and diabetics during reversed night/day circadian clocks in the time spent within target range of glucose, performance on neuro cognitive tasks, electrical brain activity, and hormonal profile.

ELIGIBILITY:
Inclusion Criteria:

* Families living in areas with high access to medical care.
* Age: 12-18 years old
* T1D diagnosis for longer than 1 year
* speaking fluent Hebrew

Exclusion Criteria:

* significant renal or liver function abnormalities
* head injuries,
* epileptic episodes
* psychiatric medications
* lack of Hebrew abilities
* disagreement to comply with all the study requests
* history of more than one episode of a severe hypoglycemic event in the past, including loss of consciousness or more than one episode of diabetic ketoacidosis.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patiets ages 12-18 years with type 1 diabetes mellitus and healthy controls same age and gender distribution
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Affects of reversal circadian clock on neuro cognitive tasks performance among healthy and T1D patients, according to glucose | 2 years
  Score of neurocognitive tests for executive function according to day/night sleeping pattern session
Affects of reversal circadian clock on Glucose Variability parameters among both healthy and T1DM adolescents . | 2 years
  Time spent in range of glucose of 70-180 mg/dl according to day/night sleeping pattern
Affects of reversal circadian clock on sleep quality among both healthy and T1DM adolescents (mainly T1DM), controlled for BMI-SDS, and mean HbA1c in T1D patients. | 2 years
  Quality of sleep according to PSQI, according to day/night sleeping pattern

SECONDARY OUTCOMES:
Melatonin profile according to night/day sleep cycle among healthy and among T1D patients | 2 years
  Differences in levels of melatonin in nmol/l between sessions and between health and T1D patients
Temperature according to night/day sleep cycle among healthy and among T1D patients | 2 years
  Differences in peripheral body temperature (celzius) between sessions and between health and T1D patients
EEG registration in accordance with the circadian curve and neurocognitive achievements | 2 years
  Power of high frequency amplitude between night/sleep sessions among T1D and healthy
MRI structural changes | 2 years
  DT1-MRI trajectoris areas of supra-chiasmatic nuclei sleeping pattern session
Hormonal profile according to night/day sleep cycle among healthy and among T1D patients | 2 years
  Differences in levels of cortisol in nmol/l between sessions and between health and T1D patients
Metabolic parameters according to night/day sleep cycle among healthy and among T1D patients | 2 years
  Differences in blood pressure (mmHG) between sessions and between health and T1D patients